CLINICAL TRIAL: NCT05710549
Title: Understanding Brain Mechanisms Involved in Autobiographical Memory Using High-density Electroencephalography and Transcranial Alternating Current Stimulation
Brief Title: Understanding Brain Mechanisms Involved in Autobiographical Memory
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lucie Bréchet (Other)
Responsible Party: Sponsor-Investigator, Lucie Bréchet, Dr., University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021-01388
Record Dates: First submitted 2023-01-12; First posted 2023-02-02 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Memory Loss
Keywords: autobiographical memory (ABM); high-density electroencephalography (EEG); magnetic resonance imaging (MRI); non-invasive brain stimulation (NIBS); transcranial alternating current stimulation (tACS)
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Memory Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- neurophysiological measurements (Experimental): 40 cognitively-unimpaired healthy young adults (age 18-35 years old), 40 cognitively-unimpaired healthy older adults (age 55+ years old), and 40 age-matched patients with mild cognitive impairment (MCI) (age 55+ years old) will be assessed using high-density electroencephalography (hdEEG) to characterize the spatiotemporal dynamics of brain oscillations during personalized, autobiographical memory (ABM) tasks.
  Interventions: Device: high-density electroencephalography (hdEEG)
- neuropsychological examination (Experimental): 40 MCI patients (age 55+ years old) will undergo 20min multi-channel protocols of transcranial alternating current stimulation; tACS (either gamma, beta, or ActiSham stimulation randomized across the three laboratory sessions) to modify cognitive functioning (MoCA score), and oscillatory brain activity during performing personalized, autobiographical memory (ABM) tasks and resting-state EEG.
  Interventions: Device: Transcranial alternating current stimulation (tACS)

INTERVENTIONS:
Device: high-density electroencephalography (hdEEG) — EEG will be recorded with a 257-channel EEG system (Geodesic Sensor Net, MegStim). An EEG net is applied at once on the head with evenly spaced sensors that provide full scalp coverage, including the cheek, Ag/Ag-Cl electrodes that are interconnected by thin rubber bands and contain small sponges soaked with saline water that touches the participant's scalp surface directly. Net application takes about 10 min to derive impedances to <30 kOhms. EEG is recorded with 1 kHz and band-pass filtered between 0.1-200 Hz. Vertex electrode Cz is used as an acquisition reference.
  Arms: neurophysiological measurements
Device: Transcranial alternating current stimulation (tACS) — tACS will be delivered by a battery-driven current stimulator Starstim SS32 (Neuroelectrics) through surface Ag/AgCl electrodes placed into holes of a neoprene cap corresponding to the international 10/20 EEG system. Gel (Parker Lab, Inc.) will be applied to optimize signal conductivity and lower impedance.
  Arms: neuropsychological examination

SUMMARY:
The overall objective of this project is to characterize the spatiotemporal dynamics of brain oscillations underpinning autobiographical memory (ABM) and the modulation of the memory network using non-invasive brain stimulation.

DETAILED DESCRIPTION:
Accumulating evidence suggests that activity in distributed networks supporting ABM is altered even decades before the expected onset of clinical symptoms in Alzheimer's disease (AD). Robust network alterations associated with age-related memory and cognitive decline have been linked to abnormal oscillatory brain rhythmic activity and functional dysconnectivity. However, the detailed neural mechanisms are still poorly understood. The investigators propose to precisely characterize the underlying neurophysiological mechanisms that lead to behavioral and cognitive disturbances in ABM of MCI patients. Specifically, hdEEG will be used to characterize the sources and spatiotemporal dynamics of the neuronal activity involved in the ABM network of 40 mild cognitive impairment (MCI) patients and compare it to 40 age-matched, older healthy participants and 40 healthy young participants. The investigators will then apply non-invasive brain stimulation in the form of transcranial alternating current stimulation (tACS) to gain novel insights into the causal role of brain oscillations in the ABM network of MCI patients.

ELIGIBILITY:
Inclusion Criteria:

Cognitively-Unimpaired Younger and Older Adults

* Age 18 to 35 years old (younger adults)
* Age 55+ years old (older adults)
* without any cognitive impairment (based on the Montreal Cognitive Assessment: MoCA)
* willing and capable to give informed consent for participation in the study after it has been thoroughly explained able
* willing to comply with all study requirements informed consent form was signed

Mild Cognitive Impairment (MCI) patients

* Age 55+ years old
* Clinical Diagnosis of MCI
* Confirmation of diagnosis will be made by the study MD based on a holistic consideration of the participant's cognitive evaluation and history
* Mini-Mental State Examination (MMSE) ≥ 18 (Mild AD ≥ 21)
* CDR ≥ .5
* Demonstration or history of autobiographical memory impairments
* On a stable dose of medications for memory loss including cholinesterase inhibitors (e.g. donepezil, rivastigmine) or memantine as defined as 6 consecutive weeks of treatment at an unchanging dose
* Minimum of completed 8th-grade education
* willing and capable to give informed consent for participation in the study after it has been thoroughly explained - note that to ensure this in the case of the MCI participants, a cut-off of MOCA score >18 will be applied
* able and willing to comply with all study requirements informed consent form was signed

Exclusion Criteria:

Cognitively-Unimpaired Younger and Older Adults

* any cognitive impairment captured by the Montreal Cognitive Assessment (MoCA) - score < 26
* major psychiatric co-morbidity including major depressive disorder, schizophrenia, or psychosis
* blindness or other disabilities that prevent task performance
* Contraindication for undergoing MRI
* Any metal in the brain or skull (excluding dental fillings) or elsewhere in the body unless cleared by the responsible covering MD (e.g. MRI compatible joint replacement)

Mild Cognitive Impairment (MCI) patients

* Age < 55 years old
* Any current diagnosis of a major psychiatric disorder (e.g., schizophrenia, bipolar disorder, major depressive disorder)
* Other than MCI, any history of other progressive or genetic neurologic disorder (e.g. Parkinson's disease, multiple sclerosis, tubular sclerosis) or acquired neurological disease (e.g. stroke, traumatic brain injury, tumor), including intracranial lesions
* History of head trauma resulting in prolonged loss of consciousness
* Current history of poorly controlled headaches including chronic medication for migraine prevention
* History of fainting spells of unknown or undetermined etiology that might constitute seizures
* History of seizures, diagnosis of epilepsy, or immediate (1st-degree relative) family history of epilepsy with the exception of a single seizure of benign etiology (e.g. febrile seizures) in the judgment of a board-certified neurologist
* Any unstable medical condition or chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.) or study complication
* contraindications to tACS, as recorded on a standardized screening questionnaire, which include a reported seizure within the past two years, use of neuroactive drugs, self-reported presence of specific implanted medical devices (e.g., deep brain stimulator, medication infusion pump, cochlear implant, pacemaker, etc.), or the presence of any active dermatological condition, such as eczema, on the scalp
* Contraindication for undergoing MRI or receiving tACS
* Any metal in the brain or skull (excluding dental fillings) or elsewhere in the body unless cleared by the responsible covering MD (e.g. MRI compatible joint replacement)
* Any devices such as a pacemaker, medication pump, nerve stimulator, TENS unit, ventriculoperitoneal shunt unless cleared by the responsible covering MD

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Spatiotemporal dynamic changes measured with electroencephalography (hdEEG) | up to 30 minutes
  Changes in spatiotemporal dynamics in different frequency bands (theta, alpha, beta, gamma) will be assessed with hdEEG
Cognitive Assessment | baseline
  The Montreal Cognitive Assessment (MOCA) will be administered to characterize the cognitive status

CONTACTS AND LOCATIONS:
Overall Officials: Lucie Bréchet, PhD, Principal Investigator — University of Geneva (UNIGE); Paul G Unschuld, Prof. MD, Study Chair — Geneva University Hospitals (HUG)
Locations (1):
- University of Geneva, Campus Biotech, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Background] Brechet L, Brunet D, Birot G, Gruetter R, Michel CM, Jorge J. Capturing the spatiotemporal dynamics of self-generated, task-initiated thoughts with EEG and fMRI. Neuroimage. 2019 Jul 1;194:82-92. doi: 10.1016/j.neuroimage.2019.03.029. Epub 2019 Mar 19. PMID 30902640
- [Background] Roehri N, Brechet L, Seeber M, Pascual-Leone A, Michel CM. Phase-Amplitude Coupling and Phase Synchronization Between Medial Temporal, Frontal and Posterior Brain Regions Support Episodic Autobiographical Memory Recall. Brain Topogr. 2022 Mar;35(2):191-206. doi: 10.1007/s10548-022-00890-4. Epub 2022 Jan 26. PMID 35080692
- [Background] Michel CM, He B. EEG source localization. Handb Clin Neurol. 2019;160:85-101. doi: 10.1016/B978-0-444-64032-1.00006-0. PMID 31277878